CLINICAL TRIAL: NCT01270646
Title: Study of the Role of Intraventricular Electrical Activation in the Treatment of Congestive Heart Failure by Cardiac Resynchronization Therapy: Invasive Evaluation and Validation of Non-Invasive Strategy Using CardioInsight ®
Brief Title: Impact of Intraventricular Electrical Activation in Resynchronization Therapy
Acronym: CARTO-CRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2010/29
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure; Cardiomyopathy, Dilated; Coronary Disease
Keywords: Cardiac insufficiency; Invasive procedure; Heart Failure; Noninvasive procedure; Congestive Heart Failure; Mapping; Cardiac resynchronisation therapy; Open study; Cardiac Pacings, Artificial; Hemodynamics
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraventricular Electrical Activation (Experimental)
  Interventions: Device: Invasive mapping with CARTO3 system and Non-Invasive mapping with CardioInsight Atlas EC Mapping system

INTERVENTIONS:
Device: Invasive mapping with CARTO3 system and Non-Invasive mapping with CardioInsight Atlas EC Mapping system — Day 1: CRT device is implanted under general anesthesia in a conventional fashion. The coronary sinus leads will be implanted guided by the acute hemodynamic response (+(dP/dt)max) using a RADI guide wire. After device implantation, a steerable mapping catheter will be inserted in the Left Ventricle (LV) cavity to build a tridimensional activation map of the LV. This map will be obtained with and without CRT. From these maps different parameters describing LV activation will be measured and compared between patients with and without CRT.
  Day 5±2: A non-invasive map of the LV will be recorded with the CardioInsight ® system with and without CRT. The same parameters will be measured and compared with those obtained with invasive mapping.

SUMMARY:
Impact of intraventricular electrical activation in resynchronization therapy. We seek to evaluate the impact of Cardiac Resynchronization Therapy (CRT) on electrical activation of the Left Ventricle (LV). The first goal of the study is to evaluate if CRT is able to decrease the heterogeneity of LV activation in heart failure patients. A second goal is to evaluate the electrical determinant of clinical response to CRT using invasive and non-invasive mapping technology.

DETAILED DESCRIPTION:
Comprehensive study, prospective, monocentric and cohort study.

Biventricular pacing is an effective therapy to improve end stage heart failure patients, however up to 30% of patients are unresponsive to this therapy. Among others, optimization of Left Ventricle (LV) pacing site location is critical to optimize response to Cardiac Resynchronization Therapy (CRT). Whether a better comprehension of baseline LV electrical activation can help to determine optimal LV lead location remains to be investigated.

After informed consent patients are included in the sudy. Day 1: CRT device is implanted under general anesthesia in a conventional fashion. The coronary sinus leads will be implanted guided by the acute hemodynamic response (+(dP/dt)max) using a RADI guide wire. After device implantation, a steerable mapping catheter will be inserted in the LV cavity to build a tridimensional activation map of the LV. This map will be obtained with and without CRT. From these maps different parameters describing LV activation will be measured and compared between patients with and without CRT. Quantitative parameters: Global LV activation time (LVATG) (primary outcome); septal activation time (LVTAS); Global intra-LV dispersion time and Qualitative parameters: presence of intraLV line of block, area of late activation. Day 5±2: A non-invasive map of the LV will be recorded with the CardioInsight ® system with and without CRT. The same parameters will be measured and compared with those obtained with invasive mapping. A 3 and 6 months follow-up visit including clinical, biological evaluation (NYHA status, 6-min walking test, BNP) of the patients will be performed with an additional transthoracic echocardiography at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 or above)
* Sinus rhythm
* Patient must have signed informed consent
* Cardiac insufficiency of whatever cause (ischemic or non-ischemic)
* Patient eligible for implantation of a ventricular resynchronization device or patient with a ventricular resynchronization device having a procedure of ventricular tachycardia ablation
* Left ventricular ejection fraction <35%
* NYHA Class II to IV with optimal medical treatment
* Patient covered by national healthcare insurance

Exclusion Criteria:

* Pregnant woman
* Sequel of transmural myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Evolution of the Global Left Ventricle activation time (LVATG) with and without Cardiac Resynchronization Therapy (CRT). | Day 1 : End of CRT device implantation

SECONDARY OUTCOMES:
Number, area and location of line of conduction block in the Left Ventricle | Day 1 : End of CRT device implantation
Area of the latest activated region of the Left Ventricle | Day 1 : End of CRT device implantation
Number, area and location of LV region activated after the end of surface QRS | Day 1 : End of CRT device implantation
Septal activation time (LVTAS) | Day 1 : End of CRT device implantation
Global intra-Left Ventricular dispersion time | Day 1 : End of CRT device implantation
Determination of the electrical parameters associated with good clinical response to CRT at 6 months. | 6 months after CRT device implantation
Non-invasive mapping: Same criteria evaluated non-invasively using CardioInsight ® with and without Cardiac Resynchronization Therapy activated. | Between 3 to 7 days after CRT device implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital cardiologique du Haut-Lévêque, Pr. Haïssaguerre's department, 3rd Floor, Pessac, France

REFERENCES:
- [Derived] Huntjens PR, Ploux S, Strik M, Walmsley J, Ritter P, Haissaguerre M, Prinzen FW, Delhaas T, Lumens J, Bordachar P. Electrical Substrates Driving Response to Cardiac Resynchronization Therapy: A Combined Clinical-Computational Evaluation. Circ Arrhythm Electrophysiol. 2018 Apr;11(4):e005647. doi: 10.1161/CIRCEP.117.005647. PMID 29654125